CLINICAL TRIAL: NCT05457322
Title: The RELAX Trial: Nonpharmaceutical Intervention for Nocturnal Muscle Cramps
Acronym: RELAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Elliot B. Tapper, Associate Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00216488
Record Dates: First submitted 2022-07-09; First posted 2022-07-14 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cramps; Muscle Cramp
Keywords: Nighttime muscle cramps; Cirrhosis; Liver disease; Qualify of life; Sleep; Non-Pharmaceutical intervention
MeSH Terms: conditions — Muscle Cramp; Fibrosis; Liver Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral intervention one (Experimental)
  Interventions: Behavioral: Behavioral intervention one
- Behavioral intervention two (Experimental)
  Interventions: Behavioral: Behavioral intervention two

INTERVENTIONS:
Behavioral: Behavioral intervention one — Participants will view or listen to audiovisual material and engage in a daily 10-minute exercise. Following the practice period participants will continue to do the true 28-day intervention period in which they were randomized to.
  Arms: Behavioral intervention one
Behavioral: Behavioral intervention two — Participants will view or listen to audiovisual material and engage in a daily 10-minute exercise. Following the practice period participants will continue to do the true 28-day intervention period in which they were randomized to.
  Arms: Behavioral intervention two

SUMMARY:
The purpose of the study is to learn about reducing the symptoms and severity of nighttime lower body muscle cramps in patients with and without cirrhosis.

Eligible participants will have an initial 7-day practice phase, followed by 28 days of one of two behavioral interventions.

DETAILED DESCRIPTION:
The interventions in this trial can be done at home. Openly discussing the intervention groups with all participants prior to randomization thus poses a high risk of tainting the study because subjects in the one group may start doing the other groups exercises after having heard about it during the consent process as a way to potentially reduce the symptoms and severity of painful muscle cramps. Therefore, this study will conceal information regarding the nature of the interventions. Only participants randomized to the true intervention group will be told during the study period what the behavioral intervention is. Additionally, the title of this trial upon registration is listed slightly differently than it is listed with the Institutional Review Board (IRB), to provide scientific integrity with the masking requirements. When the trial is completed, the title will be amended to match the IRB approved title. At the conclusion of the study, at the time of the final follow-up assessments, all participants will be debriefed on the use of the concealment of the study object in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants have painful muscle spasms, cramps, or charley horses at night in feet or legs.
* Participants have muscle cramps that happen at least four times in the past month. And the muscle cramps bother them.
* For Cirrhosis patients only: diagnosis of cirrhosis based upon:

  1. liver biopsy, or
  2. history of cirrhosis complication: ascites, variceal bleeding, hepatic encephalopathy, or
  3. 2 of the following 4 criteria:
* Ultrasound (US), computerized tomography (CT) or Magnetic resonance imaging (MRI) imaging findings of cirrhosis (cirrhotic appearing liver, splenomegaly, varices, ascites)
* FibroScan liver stiffness score >13 kilopascal (kPa)
* Laboratory testing: aspartate aminotransferase (AST)/platelet ratio index (APRI) >2.0
* CT, MRI or esophagogastroduodenoscopy (EGD) showing presence of esophageal varices

Exclusion Criteria:

* Non-English speaking
* Unable or unwilling to provide consent
* Pregnancy via self-report
* Disorientation at the time of enrollment
* History of multiple sclerosis
* History of cerebral palsy
* History of stroke with paralysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Change in cramp severity after 35-days as measured by the Visual Analog Scale for Cramps | baseline, 35 days
  This is a one question scale from 0 to 10; 0 indicates no cramps and 10 indicates worst cramps imaginable.

SECONDARY OUTCOMES:
Patient global impression of change (PGIC) | 35 days
  This is a one question survey in which the participants rate overall status as one of the following:
  Very Much Improved, Much Improved, Minimally Improved, No Change, Minimally Worse, Much Worse, Very Much Worse. Comparison of PGIC scores at 35 days between both arms.
Change in sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI). | baseline, 35 days
  This is a one question survey in which the participants rate overall sleep quality as one of the following: Very good, Good, Fair, Bad, Very bad.

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Tapper, MD, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - Cedars-Sinai, Los Angeles, California
  - University of Miami Health System, Miami, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Baylor, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No